CLINICAL TRIAL: NCT01128348
Title: A Patient Advocate and Literacy-Based Treatment of Asthma
Acronym: HAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Andrea Apter, Professor of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 700; RC1HL099612 (NIH)
Record Dates: First submitted 2010-05-20; First posted 2010-05-21 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Asthma
Keywords: asthma; adherence; quality of life; health literacy; health disparities
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- patient advocate (Experimental): Patient advocate works with patient before, during, and after a visit to asthma doctor.
  Patient receives video of asthma education materials
  Interventions: Behavioral: patient advocate
- asthma education (Active Comparator): Patient receives video of asthma education materials
  Interventions: Behavioral: patient advocate

INTERVENTIONS:
Behavioral: patient advocate — patient advocate works with patient to navigate practice and social barriers and to facilitate patient-provider communication

SUMMARY:
Half of US adults have no more than basic reading and numerical skills. A consequence is inadequate health literacy, which is associated with unsatisfactory patient-provider communication and poor health outcomes in chronic diseases, including asthma. We have adapted a patient navigator intervention to address asthma in high risk communities as a practical, immediate, and sustainable method of achieving effective health literacy in patients low health literacy. This intervention will lead to improved adherence and asthma control, attenuating health disparities so marked in asthma. It is compared for efficacy and cost-effectiveness with asthma education.

DETAILED DESCRIPTION:
This application addresses broad Challenge Area (05), Comparative Effectiveness Research, and Specific Challenge Topic 05-MD105, Health Literacy. Half of US adults have no more than basic reading and numerical skills; inadequate health literacy is a consequence. It is associated with unsatisfactory patient-provider communication and poor health outcomes in chronic diseases including asthma. We found low numeracy to be associated with prior ED visits and hospitalizations for asthma and determined that numerical skill may attenuate the association of minority status with lower asthma-related quality of life. We propose a Patient Advocate Intervention (PAI) as the most practical immediate but sustainable method of achieving effective health literacy (EHL) (understanding of asthma management and the practice/health system). Adapted from the Patient Navigator of Harold P. Freeman, MD and informed by focus groups of asthma patients, the PAI addresses low literacy, facilitating patient-provider communication surrounding self-management and navigation of the practice and health system to ensure medical recommendations can be accomplished. The PA is a nonprofessional with guidance from a social worker who will assist with and model preparations for a visit with the asthma doctor, attend the visit, and afterwards confirm understanding as well as facilitate scheduling, obtaining insurance coverage, and overcoming other barriers to carrying out medical advice. The primary outcome is electronically-monitored use of inhaled corticosteroids (ICS), the treatment of choice for all but the mildest asthma. ICS use is a marker of successful patient-provider communication. Other outcomes are asthma-related: hospitalizations, ED visits, change in FEV1, and asthma-related quality of life. We hypothesize that the PAI will improve these outcomes by promoting EHL.

We will enroll 84 adults with a high prevalence of low numerical skills who are approximately 67% black and 10% Latino with moderate or severe asthma to carry out the following Specific Aims. Specific Aim 1: refine and evaluate the feasibility of PAI and Specific Aim 2: conduct a randomized comparison of PAI with standard asthma education to obtain effect size estimates for ICS adherence and asthma-related outcomes for a future R01 confirmatory randomized trial of the final version of PAI. Exploratory analyses will assess EHL as a mediator, various moderators, and estimate the incremental costs of PAI. This novel project fills several research gaps. It 1) compares and tests an intervention addressing literacy to improve health, one that can easily be incorporated into practice to better patient self-management and preventive care, 2) is a potentially long-lasting intervention which will benefit all patients, especially those with low health literacy, and 3) will potentially improve prevention of asthma exacerbations, reducing the need for ED use.

ELIGIBILITY:
Inclusion Criteria:

* physician's diagnosis of asthma
* prescribed inhaled steroid
* moderate or severe asthma according to NHLBI Guidelines
* evidence of reversible airflow obstruction and improvement with bronchodilator
* Did not participate in the experimental arm (problem-solving) of WIN Study, HL073932

Exclusion Criteria:

* significant other current pulmonary or cardiac disease
* severe psychiatric problems making it impossible to understand or carryout the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
adherence to prescribed inhaled corticosteroid regimen | 16 weeks

SECONDARY OUTCOMES:
change in FEV1 | 16 weeks
asthma-related quality of life | 16 weeks
asthma control | 16 weeks
emergency department visits for asthma | 16 weeks
hospitalizations for asthma | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andrea J Apter, MD, MSc, MA, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Black HL, Priolo C, Gonzalez R, Geer S, Adam B, Apter AJ. An analysis of contextual information relevant to medical care unexpectedly volunteered to researchers by asthma patients. J Asthma. 2012 Sep;49(7):731-7. doi: 10.3109/02770903.2012.699988. Epub 2012 Jul 13. PMID 22788543
- [Background] Black HL, Priolo C, Akinyemi D, Gonzalez R, Jackson DS, Garcia L, George M, Apter AJ. Clearing clinical barriers: enhancing social support using a patient navigator for asthma care. J Asthma. 2010 Oct;47(8):913-9. doi: 10.3109/02770903.2010.506681. PMID 20846085
- [Background] Krishnan JA, Schatz M, Apter AJ. A call for action: Comparative effectiveness research in asthma. J Allergy Clin Immunol. 2011 Jan;127(1):123-7. doi: 10.1016/j.jaci.2010.08.032. Epub 2010 Sep 19. PMID 20855111
- [Background] Apter AJ, Wang X, Bogen DK, Rand CS, McElligott S, Polsky D, Gonzalez R, Priolo C, Adam B, Geer S, Ten Have T. Problem solving to improve adherence and asthma outcomes in urban adults with moderate or severe asthma: a randomized controlled trial. J Allergy Clin Immunol. 2011 Sep;128(3):516-23.e1-5. doi: 10.1016/j.jaci.2011.05.010. Epub 2011 Jun 25. PMID 21704360